CLINICAL TRIAL: NCT03614676
Title: A Prospective Epidemiological Study of Pregnancy Outcomes and of Events of Interest in Pregnant Women, Neonates and Infants (PEPNI)
Brief Title: A Study of Outcomes and Events of Interest in Pregnant Women, Neonates and Infants and of RSV Surveillance
Acronym: PEPNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 207636
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: third trimester; Respiratory Syncytial Virus (RSV) illness; Pregnancy; Maternal Immunization; Pregnant Women; Neonates; Respiratory Tract Illness
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Single Group Assignment is selected because this is a low-interventional, epidemiological study. As such, the study does not have multiple groups/treatment arms that will be compared against one another statistically in the way two study arms would be compared against each other in a clinical trial. Instead, the study will longitudinally follow pregnant women through a 42-day post-delivery period and will also follow the infants born to these women. It should be noted that these are the two populations listed in the protocol, but these are not two groups that will compared against one another. Statistical analyses will be conducted within each group and some analyses will be done across the two groups. However, these two groups should not be considered equivalent to two study arms. This explains why a single group assignment is appropriate while two study groups (mothers and infants) will be examined.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant Women/Mothers Group (Other): Subjects, 18 to 45 years of age enrolled in the study in view of determining pregnancy outcomes and related events of interest, as well as the occurrence of lower respiratory tract illness (LRTI) associated with respiratory syncytial virus (RSV).
  Interventions: Procedure: Blood sample collection; Procedure: Cord blood sample collection; Other: Maternal Diary Card
- Neonates/Infants Group (Other): Infants born to mothers aged 18-45 years old, enrolled for the collection of infant events of interest, nasal swabs and the incidence of RSV LRTI and RSV hospitalization.
  Interventions: Procedure: Nasal Swab collection; Other: Infant Diary Card

INTERVENTIONS:
Procedure: Blood sample collection — Venous blood samples will be collected from the maternal subjects at Day 1 and Day 56 of the study and at delivery.
  Arms: Pregnant Women/Mothers Group
Procedure: Cord blood sample collection — Collection of cord blood samples from maternal subjects will occur, at delivery
  Arms: Pregnant Women/Mothers Group
Other: Maternal Diary Card — Completion of Diary Card about health by pregnant woman/ mother, from enrolment through week 6 post delivery.
  Arms: Pregnant Women/Mothers Group
Procedure: Nasal Swab collection — Collection of nasal swabs from infants with potential LRTIs, from birth to 12 months of age.
  Arms: Neonates/Infants Group
Other: Infant Diary Card — Completion of Diary Card about health of infant from birth to 12 months of age.
  Arms: Neonates/Infants Group

SUMMARY:
The purpose of this study is to assess pregnancy outcomes, and maternal, as well as neonatal events of interest in healthy pregnant women and their new-borns. The study will also determine incidence of lower respiratory tract illness (LRTI) caused by respiratory syncytial virus (RSV) in the new-borns during their first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women 18-45years of age who are ≥ 24 0/7 weeks GA at screening and ≤ 27 6/7 weeks GA at Visit 1, as established by ultrasound examination and/or last menstrual period (LMP) date
* Women with pre-pregnancy body mass index (BMI) ≥18.5 and ≤ 39.9 kg/m2.
* Women whose pregnancy is considered low risk, based on medical history, obstetric history, and clinical findings during the current pregnancy
* Women who had no significant findings (such as abnormal fetal morphology, amniotic fluid levels, placenta, or umbilical cord) observed during a Level 2 ultrasound (fetal morphology assessment).
* Human Immunodeficiency Virus (HIV) uninfected women who have been tested within the past year and have documented HIV negative test results.
* Individuals who give written or witnessed/thumb printed informed consent after the study has been explained according to local regulatory requirements.

  * The informed consent given at screening should either include consent for both the mother's participation and participation of the infant after the infant's birth (if consistent with local regulations/guidelines), or consent for the mother's participation and expressed willingness to consider permitting the infant to take part after the infant has been born (if local regulations/guidelines require parent(s) to provide an additional informed consent after the infant's birth).
  * Both mother and father should consent if local regulations/guidelines require it.
* Individuals who consent to have cord blood collected at delivery for the purpose of the study;
* Individuals who plan to reside in the study area for at least one year after delivery.
* Individuals who are in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
* Individuals who, in the opinion of the investigator can and will comprehend and comply with all study procedures
* Infants who were in utero at the time maternal (and paternal, if required) informed consent was given, and who are live-born.
* If local law requires it: Written or witnessed/thumb printed informed consent for study participation of the infant obtained from parent(s)/Legally Accepted Representative [LAR(s)] within 21 days of birth.

Exclusion Criteria:

* Individuals determined to have one of the following conditions associated with increased risk for a serious obstetrical complication

  * Gestational hypertension;
  * Gestational diabetes uncontrolled by diet and exercise;
  * Pre-eclampsia or eclampsia;
  * Multiple pregnancy;
  * Intrauterine growth restriction;
  * Placenta previa;
  * Polyhydramnios;
  * Oligohydramnios;
* Individuals determined to have (during the current pregnancy) one of the following infections or conditions associated with risk of adverse outcome:

  * Known or suspected:

    * Syphilis infection,
    * Parvovirus B19,
    * Rubella infection,
    * primary herpes simplex infection,
    * primary cytomegalovirus infection,
    * varicella infection,
    * Zika infection,
    * Active tuberculosis infection,
  * Incompetent cervix or cerclage
* Individuals who have any underlying condition or infection that would predispose them to increased risk for a serious obstetrical complication that is not mentioned above
* Individuals who have behavioural or cognitive impairment or psychiatric disease that, in the opinion of the investigator, could interfere with the subject's ability to participate in the study;
* Individuals who have known or suspected impairment of the immune system, an active autoimmune disorder that is not well-controlled, or who are receiving systemic immunosuppressive therapy;
* Individuals participating in any concurrent clinical trial during the current pregnancy;
* Individuals pregnant with a fetus with a confirmed or suspected major congenital anomaly at the time of enrolment.
* Child in care

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4493 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Argentina (4):
  - GSK Investigational Site, Villanueva- Guaymallen, Mendoza Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Río Cuarto
- GSK Investigational Site, Dhaka, Bangladesh
- Brazil (3):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Santa Maria, Rio Grande do Sul
  - GSK Investigational Site, Ribeirão Preto, São Paulo
- Colombia (4):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Medellín
  - GSK Investigational Site, Villavicencio
- Malaysia (4):
  - GSK Investigational Site, Alor Star
  - GSK Investigational Site, Kota Kinabalu
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuching
- Mexico (3):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Oaxaca City
- Panama (4):
  - GSK Investigational Site, Chiriquí
  - GSK Investigational Site, Juán Diaz
  - GSK Investigational Site, La Chorrera
  - GSK Investigational Site, Panama City
- Philippines (2):
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Manila
- South Africa (3):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Parow Valley
  - GSK Investigational Site, Soshanguve
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data sets Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tullio AN, Yanni E, Coutinho CM, Sivapatham L, Lee CMF, Pallem S, Pu Y, Akawung A, Kim JH, Henry O, Mussi-Pinhata MM, Ahmed K, Del Carmen Flores Acosta C, Reyes O, Abadia de Regalado I, Arias Fernandez DA, Aurpibul L, Taher SW, Caccavo J, Ceballos A, Pichailuck C, D'Andrea Nores U, De Leon T, De Bernardi M, Dieser P, D'Silva EC, Falaschi A, Fry S, Gentile A, Teo IH, Kotze S, Lopez-Medina E, Luca R, Lucion MF, Mantaring JBIV, Marin B, Moelo M, Pinto J, Puthanakit T, Roa MF, Rodriguez Brieschke MT, Rodriguez CE, Rodriguez Nino JN, Schwarzbold AV, Sierra Garcia A, Soon R, Tinoco JC, Velasquez Penagos JA, Zaman K, Dos Santos G. A multicountry study to establish rates for pregnancy and neonatal outcomes in low- and middle-income regions. BMC Pregnancy Childbirth. 2026 Jan 14. doi: 10.1186/s12884-025-08012-1. Online ahead of print. PMID 41535781
- [Derived] Fry S, Chokephaibulkit K, Pallem S, Henry O, Pu Y, Akawung A, Kim JH, Yanni E, Tullio AN, Aurpibul L, Lee CMF, Ceballos A, Zaman K, Abadia de Regalado I, Ahmed K, Arias Fernandez DA, Taher SW, Caccavo J, Coutinho CM, D'Andrea Nores U, De Leon T, D'Silva EC, De Bernardi M, Dieser P, Falaschi A, Flores Acosta CDC, Gentile A, Teo IH, Kotze S, Lopez-Medina E, Luca R, Lucion MF, Mantaring JBIV, Marin B, Moelo M, Mussi-Pinhata MM, Pinto J, Puthanakit T, Reyes O, Roa MF, Rodriguez Brieschke MT, Rodriguez CE, Rodriguez Nino JN, Schwarzbold AV, Sierra Garcia A, Sivapatham L, Soon R, Tinoco JC, Velasquez Penagos JA, Dos Santos G. Incidence of Respiratory Syncytial Virus-Associated Lower Respiratory Tract Illness in Infants in Low- and Middle-Income Regions During the Coronavirus Disease 2019 Pandemic. Open Forum Infect Dis. 2023 Dec 1;10(12):ofad553. doi: 10.1093/ofid/ofad553. eCollection 2023 Dec. PMID 38088983

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 4493 subjects enrolled, data was not collected for one enrolled infant subject. This infant subject was therefore excluded from the study analysis. Deaths reported in the all-cause mortality module include neonatal deaths, infant deaths and maternal deaths, while deaths reported in the participant flow include only infant deaths.
Period: Overall Study
Arm/Group | Pregnant Women/Mothers Group | Neonates/Infants Group
Started | 2311 | 2181
Completed | 2195 | 2017
Not Completed | 116 | 164
Not completed — Delivery before planned visit | 2 | 0
Not completed — Consent withdrawal, not due to SAE related to study or a pregnancy related event of special interest | 34 | 0
Not completed — Migrated / moved from the study area | 30 | 22
Not completed — Lost to Follow-up | 17 | 42
Not completed — Not willing/ not able to participate in this visit | 17 | 16
Not completed — Other | 16 | 47
Not completed — Protocol Violation | 0 | 2
Not completed — Neonatal event of interest | 0 | 6
Not completed — Death in infant greater than 28 days old | 0 | 12
Not completed — Consent withdrawal not due to SAE related to study or neonatal event of special interest | 0 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Women/Mothers Group | Neonates/Infants Group | Total
Number analyzed (Participants) | 2311 | 2181 | 4492
Age, Customized [Count of Participants; unit: Participants]
  18-34 years | 1994 | 0 | 1994
  35-39 years | 262 | 0 | 262
  >=40 years | 55 | 0 | 55
  0-1 year | 0 | 2181 | 2181
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2311 | 1049 | 3360
  Male | 0 | 1132 | 1132
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity analysis was performed only for Pregnant Women/Mothers Group.
  Participants
    African Heritage/ African American: number analyzed (Participants) | 2311 | 0 | 2311
    African Heritage/ African American | 378 |  | 378
    American Indian or Alaska Native: number analyzed (Participants) | 2311 | 0 | 2311
    American Indian or Alaska Native | 51 |  | 51
    Asian-Central/South Asian Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    Asian-Central/South Asian Heritage | 214 |  | 214
    Asian-East Asian Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    Asian-East Asian Heritage | 11 |  | 11
    Asian-Japanese Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    Asian-Japanese Heritage | 1 |  | 1
    Asian-South East Asian Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    Asian-South East Asian Heritage | 693 |  | 693
    White-Arabic/North African Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    White-Arabic/North African Heritage | 48 |  | 48
    White-Caucasian/ European Heritage: number analyzed (Participants) | 2311 | 0 | 2311
    White-Caucasian/ European Heritage | 360 |  | 360
    Other - Not specified | 555 | 2181 | 2736

OUTCOME MEASURES:

1. Primary Outcome: Number of Maternal Subjects With Pregnancy Outcomes
Description: Pregnancy outcomes included: live birth with no congenital anomalies, live birth with congenital anomalies, fetal death/stillbirth loss at or after 22 weeks of gestation (antepartum stillbirth, Intrapartum stillbirth) with no congenital anomalies, fetal death/still birth loss at or after 22 weeks of gestation (antepartum stillbirth, Intrapartum stillbirth) with congenital anomalies, elective/therapeutic termination with no congenital anomalies, elective/therapeutic termination with congenital anomalies.
Time Frame: From Day 1 up to Day 42 post delivery
Population: The analysis was performed on the maternal Per Protocol Set (PPS) which included all pregnant women (mothers) meeting all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women/Mothers Group
Number analyzed (Participants) | 2222
Participants
  Live birth with no congenital anomalies | 2088
  Live birth with congenital anomalies | 18
  Antepartum fetal death/still birth with no congenital anomalies | 8
  Intrapartum fetal death/still birth with no congenital anomalies | 5
  Antepartum fetal death/still birth with congenital anomalies | 0
  Intrapartum fetal death/still birth with congenital anomalies | 1
  Elective/therapeutic termination with no congenital anomalies | 11
  Elective/therapeutic termination with congenital anomalies | 1

2. Primary Outcome: Number of Maternal Subjects With Pregnancy Related Events of Interest
Description: Pregnancy related events of interest included: maternal death, hypertensive disorders of pregnancy including gestational hypertension, pre-eclampsia and pre-eclampsia with severe features (including eclampsia), antenatal bleeding (morbidly adherent placenta, placental abruption, Caesarean scar pregnancy, uterine rupture), postpartum haemorrhage, fetal growth restriction, dysfunctional labor (first stage of labor, second stage of labor), gestational diabetes mellitus, non-reassuring fetal status, pathways to preterm birth including premature preterm rupture of membranes, preterm labour, and provider initiated preterm birth, chorioamnionitis, oligohydramnios, polyhydramnios, gestational liver disease (intrahepatic cholestasis of pregnancy [ICP], acute fatty liver of pregnancy), and maternal sepsis.
Time Frame: From Day 1 up to Day 42 post-delivery
Population: The analysis was performed on the maternal PPS which included all pregnant women (mothers) meeting all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women/Mothers Group
Number analyzed (Participants) | 2222
Participants
  Maternal death | 1
  Gestational hypertension | 72
  Pre-eclampsia | 37
  Pre-eclampsia with severe features | 16
  Morbidly adherent placenta | 1
  Placental abruption | 10
  Caesarean scar pregnancy | 0
  Uterine rupture | 0
  Postpartum haemorrhage | 37
  Fetal growth restriction | 19
  First stage of labor | 49
  Second stage of labor | 31
  Gestational diabetes mellitus | 58
  Non-reassuring fetal status | 137
  Preterm rupture of membranes | 40
  Preterm labor | 101
  Provider-initiated preterm birth | 25
  Chorioamnionitis | 13
  Oligohydramnios | 42
  Polyhydramnios | 9
  Intrahepatic Cholestatis of Pregnancy (ICP) | 3
  Acute Fatty Liver of Pregnancy | 0
  Maternal Sepsis | 0

3. Primary Outcome: Number of Infant Subjects With Neonatal Events of Interest
Description: Neonatal events of interest included: small for gestational age, low birth weight including very low birth weight, neonatal encephalopathy, congenital microcephaly (postnatally diagnosed, prenatally diagnosed), congenital anomalies [CA] (major external structural defects, internal structural defects, functional defects), neonatal death (neonatal death in a preterm live birth [gestational age greater than or equal to (≥) 28 to less than (<) 37 weeks], neonatal death in a term live birth), neonatal infections, (blood stream infections, meningitis, respiratory infection), respiratory distress in the neonate, preterm birth, failure to thrive, large for gestational age, macrosomia, any other neonatal event considered by the investigator to be of concern (e.g. neurodevelopmental delay).
Time Frame: From birth up to Day 28 post-birth
Population: The analysis was performed on the infant PPS which included all neonates/infants who born to pregnant women in the maternal PPS, meeting all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up), who have at least one time point evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates/Infants Group
Number analyzed (Participants) | 2094
Participants
  Small for gestational age | 111
  Low birth weight including very low birth weight | 156
  Neonatal encephalopathy | 6
  Congenital microcephaly-Postnatally diagnosed | 16
  Congenital microcephaly-Prenatally diagnosed | 1
  CA -Major external structural defects | 38
  CA -Internal structural defects | 46
  CA -Functional defects | 19
  Neonatal death in a preterm live birth | 3
  Neonatal death in a term live birth | 7
  Blood stream infections | 33
  Meningitis | 0
  Respiratory infection | 36
  Respiratory distress in the neonate | 94
  Preterm birth | 141
  Failure to thrive | 7
  Large for gestational age | 54
  Macrosomia | 53
  Other neonatal event considered to be of concern | 213

4. Secondary Outcome: Number of Maternal Subjects With Pregnancy Related Events of Interest for Each Global Alignment of Immunization Safety Assessment (GAIA) Level of Diagnostic Certainty
Description: Pregnancy related events of interest by GAIA level (Lv.) of diagnostic certainty (where applicable/feasible) range from Level 1 to Level 2 or 3 (Highest level of diagnostic certainty (1) to lowest level of diagnostic certainty (2 or 3)): maternal death, hypertensive disorders of pregnancy including gestational hypertension, pre-eclampsia and Pre-eclampsia with severe features (including eclampsia), antenatal bleeding (morbidly adherent placenta, placental abruption, Cesarean scar pregnancy, uterine rupture), postpartum haemorrhage, fetal growth restriction, dysfunctional labor, (first stage of labor, second stage of labor), gestational diabetes mellitus, non-reassuring fetal status, pathways to preterm birth including premature preterm rupture of membranes, preterm labour, and provider initiated preterm birth.
Time Frame: From Day 1 up to Day 42 post-delivery
Population: The analysis was performed on the maternal Per Protocol Set (PPS) which includes all pregnant women (mothers) meeting all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women/Mothers Group
Number analyzed (Participants) | 2222
Participants
  Maternal death-Lv.1 | 0
  Maternal death-Lv. 2 | 0
  Maternal death-Lv. 3 | 1
  Gestational hypertension-Lv. 1 | 27
  Gestational hypertension-Lv. 2 | 23
  Pre-eclampsia-Lv. 1 | 17
  Pre-eclampsia-Lv. 2 | 12
  Pre-eclampsia with severe features-Lv. 1 | 13
  Pre-eclampsia with severe features-Lv. 2 | 0
  Morbidly adherent placenta-Lv. 1 | 0
  Morbidly adherent placenta-Lv. 2 | 1
  Placental abruption-Lv. 1 | 3
  Placental abruption-Lv. 2 | 4
  Caesarean scar pregnancy-Lv. 1 | 0
  Caesarean scar pregnancy-Lv. 2 | 0
  Uterine rupture-Lv. 1 | 0
  Uterine rupture-Lv. 2 | 0
  Postpartum haemorrhage-Lv. 1 | 5
  Postpartum haemorrhage-Lv. 2 | 17
  Postpartum haemorrhage-Lv. 3 | 6
  Fetal growth restriction-Lv. 1a | 5
  Fetal growth restriction-Lv. 2a | 2
  Fetal growth restriction-Lv. 1b | 2
  Fetal growth restriction-Lv. 2b | 7
  Dysfunctional labor: First stage of labor-Lv. 1 | 34
  Dysfunctional labor: First stage of labor-Lv. 2 | 9
  Dysfunctional labor: Second stage of labor-Lv. 1 | 17
  Dysfunctional labor: Second stage of labor-Lv. 2 | 10
  Gestational diabetes mellitus-Lv. 1 | 43
  Gestational diabetes mellitus-Lv. 2 | 3
  Gestational diabetes mellitus-Lv. 3 | 11
  Non-reassuring fetal status-Lv. 1 | 26
  Non-reassuring fetal status-Lv. 2 | 17
  Non-reassuring fetal status-Lv. 3 | 30
  Preterm rupture of membranes-Lv. 1 | 14
  Preterm rupture of membranes-Lv. 2 | 7
  Preterm rupture of membranes-Lv. 3 | 13
  Preterm labor-Lv. 1 | 29
  Preterm labor-Lv. 2 | 16
  Preterm labor-Lv. 3 | 14
  Provider-initiated preterm birth-Lv. 1 | 23
  Provider-initiated preterm birth-Lv. 2 | 1
  Provider-initiated preterm birth-Lv. 3 | 1

5. Secondary Outcome: Number of Infant Subjects With Neonatal Events of Interest for Each GAIA Level of Diagnostic Certainty
Description: Neonatal events of interest by GAIA level (Lv.) of diagnostic certainty, range from Level 1 to Level 4 or 5 (Highest level of diagnostic certainty (1) to lowest level of diagnostic certainty (4 or 5 based on the neonatal events)): small for gestational age, low birth weight including very low birth weight, neonatal encephalopathy, congenital microcephaly (postnatally diagnosed, prenatally diagnosed), congenital anomalies [CA] (major external structural defects, internal structural defects, functional defects), neonatal death (neonatal death in a preterm live birth [gestational age ≥ 28 to <37 weeks], neonatal death in a term live birth), neonatal infections (blood stream infections, meningitis, respiratory infection, respiratory distress in the neonate, preterm birth, failure to thrive, large for gestational age, macrosomia, any other neonatal event considered by the investigator to be of concern (e.g. neurodevelopmental delay).
Time Frame: From birth through Day 28 of life
Population: The analysis was performed on the infant PPS which included all neonates/infants meeting all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up), who have at least one time point evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates/Infants Group
Number analyzed (Participants) | 2094
Participants
  Small for gestational age-Lv. 1 | 46
  Small for gestational age-Lv. 2a | 28
  Small for gestational age-Lv. 2b | 11
  Small for gestational age-Lv. 3a | 2
  Small for gestational age-Lv. 3b | 2
  Small for gestational age-Lv. 4 | 0
  Low birth weight including very low weight-Lv. 1 | 106
  Low birth weight including very low weight-Lv. 2 | 11
  Low birth weight including very low weight-Lv. 3 | 16
  Low birth weight including very low weight-Lv. 4 | 5
  Neonatal encephalopathy-Lv. 1 | 4
  Neonatal encephalopathy-Lv. 2 | 0
  Neonatal encephalopathy-Lv. 3 | 2
  Congenital microcephaly postnat. diagnosed-Lv. 1 | 7
  Congenital microcephaly postnat. diagnosed-Lv. 2a | 3
  Congenital microcephaly postnat. diagnosed-Lv. 2b | 4
  Congenital microcephaly postnat. diagnosed-Lv. 3a | 0
  Congenital microcephaly postnat. diagnosed-Lv. 3b | 0
  Congenital microcephaly postnat. diagnosed-Lv. 4 | 0
  Congenital microcephaly prenat. diagnosed-Lv. 1a | 0
  Congenital microcephaly prenat. diagnosed-Lv. 1b | 0
  Congenital microcephaly prenat. diagnosed-Lv. 2 | 0
  Congenital microcephaly prenat. diagnosed-Lv. 3a | 0
  Congenital microcephaly prenat. diagnosed-Lv. 3b | 0
  Congenital microcephaly prenat. diagnosed-Lv. 4 | 0
  CA- Major external structural defects-Lv. 1 | 9
  CA- Major external structural defects-Lv. 2 | 5
  CA- Major external structural defects-Lv. 3 | 3
  CA- Major external structural defects-Lv. 4 | 0
  CA- Internal structural defects-Lv. 1 | 12
  CA- Internal structural defects-Lv. 2 | 9
  CA- Internal structural defects-Lv. 3 | 22
  CA- Internal structural defects-Lv. 4 | 0
  CA- Functional defects-Lv. 1 | 14
  CA- Functional defects-Lv. 2 | 3
  CA- Functional defects-Lv. 3 | 0
  CA- Functional defects-Lv. 4 | 1
  Neonatal death in a preterm live birth-Lv. 1 | 2
  Neonatal death in a preterm live birth-Lv. 2 | 1
  Neonatal death in a preterm live birth-Lv. 3 | 0
  Neonatal death in a term live birth-Lv. 1 | 3
  Neonatal death in a term live birth-Lv. 2 | 3
  Neonatal death in a term live birth-Lv. 3 | 0
  Blood stream infections-Lv. 1 | 7
  Blood stream infections-Lv. 2 | 9
  Blood stream infections-Lv. 3 | 6
  Meningitis-Lv. 1 | 0
  Meningitis-Lv. 2 | 0
  Meningitis-Lv. 3a | 0
  Meningitis-Lv. 3b | 0
  Respiratory infection-Lv. 1 | 3
  Respiratory infection-Lv. 2 | 9
  Respiratory infection-Lv. 3 | 13
  Respiratory distress in the neonate-Lv. 1 | 59
  Respiratory distress in the neonate-Lv. 2 | 14
  Respiratory distress in the neonate-Lv. 3 | 2
  Respiratory distress in the neonate-Lv. 4 | 11
  Respiratory distress in the neonate-Lv. 5 | 0
  Preterm birth-Lv. 1 | 73
  Preterm birth-Lv. 2a | 43
  Preterm birth-Lv. 2b | 19
  Preterm birth-Lv. 3a | 2
  Preterm birth-Lv. 3b | 1
  Failure to thrive-Lv. 1 | 4
  Failure to thrive-Lv. 2a | 0
  Failure to thrive-Lv. 2v | 0
  Failure to thrive-Lv. 3a | 0
  Failure to thrive-Lv. 3b | 0

6. Secondary Outcome: Respiratory Syncytial Virus Type A (RSV-A) Neutralizing Antibody Titers in Maternal Blood
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were expressed Geometric Mean Titers (GMT) with 95% Confidence Interval (CI) in Estimated Dilution 60 (ED60) and were measured on blood samples collected from vaccinated maternal subjects.
Time Frame: At delivery
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pregnant Women/Mothers Group
Number analyzed (Participants) | 2012
Titers | 547.6 [530.0 to 565.8]

7. Secondary Outcome: RSV-A Neutralizing Antibodies Titers in Cord Blood
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. The corresponding antibody titers were presented as GMTs, expressed in ED60. The antibodies were measured on the cord blood sample collected at delivery.
Time Frame: At delivery
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pregnant Women/Mothers Group
Number analyzed (Participants) | 1886
Titers | 751.5 [724.7 to 779.4]

8. Secondary Outcome: Incidence Rates of RSV Lower Respiratory Tract Infection (LRTI) or Severe LRTI or Very Severe LRTI for Infant Subjects as Defined by the LRTI Case Definition
Description: The incidence rate was calculated by dividing the number of infant subjects reporting first episodes over the follow-up period, to the total person-years. LRTI Case definition by WHO (Modjarrad, 2016): LRTI is diagnosed when infant has history of cough OR difficulty in breathing AND SpO2 < 95%, OR RR increase AND Confirmed RSV infection. Severe LRTI is diagnosed when an infant with RSV LRTI has oxygen saturation <93% or lower chest wall drawing. Very severe LRTI is diagnosed when an infant with RSV LRTI has oxygen saturation <90%, OR inability to feed OR failure to respond / unconscious.
Time Frame: From birth up to 1 year of age
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Neonates/Infants Group
Number analyzed (Participants) | 2094
Cases per 100 person-years
  0 months | 0 [0 to 2.1]
  1 month: number analyzed (Participants) | 2081
  1 month | 2.3 [0.6 to 6.0]
  2 months: number analyzed (Participants) | 2070
  2 months | 0.6 [0 to 3.2]
  3 months: number analyzed (Participants) | 2064
  3 months | 0 [0 to 2.1]
  4 months: number analyzed (Participants) | 2061
  4 months | 0.6 [0 to 3.2]
  5 months: number analyzed (Participants) | 2054
  5 months | 1.2 [0.1 to 4.2]
  6 months: number analyzed (Participants) | 2047
  6 months | 1.8 [0.4 to 5.1]
  7 months: number analyzed (Participants) | 2043
  7 months | 3.5 [1.3 to 7.7]
  8 months: number analyzed (Participants) | 2038
  8 months | 3.6 [1.3 to 7.8]
  9 months: number analyzed (Participants) | 2033
  9 months | 3.6 [1.3 to 7.8]
  10 months: number analyzed (Participants) | 2032
  10 months | 1.2 [0.1 to 4.3]
  11 months: number analyzed (Participants) | 2025
  11 months | 0.7 [0 to 3.7]

9. Secondary Outcome: Incidence Rates of Infant Subjects With RSV Hospitalizations
Description: The incidence rate was calculated by dividing the number of subjects reporting first episodes over the follow-up period to the total person-years. RSV hospitalizations definition by WHO (Modjarrad, 2015): Infant has confirmed RSV infection AND hospitalized for acute medical condition.
Time Frame: From birth up to 1 year of age
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cases per 100 person-years
Arm/Group | Neonates/Infants Group
Number analyzed (Participants) | 2094
Cases per 100 person-years
  0 months | 0.6 [0 to 3.2]
  1 month: number analyzed (Participants) | 2081
  1 month | 0.6 [0 to 3.2]
  2 months: number analyzed (Participants) | 2070
  2 months | 0 [0 to 2.1]
  3 months: number analyzed (Participants) | 2064
  3 months | 0 [0 to 2.1]
  4 months: number analyzed (Participants) | 2061
  4 months | 0.6 [0 to 3.2]
  5 months: number analyzed (Participants) | 2054
  5 months | 0.6 [0 to 3.3]
  6 months: number analyzed (Participants) | 2047
  6 months | 0 [0 to 2.2]
  7 months: number analyzed (Participants) | 2043
  7 months | 0 [0 to 2.2]
  8 months: number analyzed (Participants) | 2038
  8 months | 0.6 [0 to 3.3]
  9 months: number analyzed (Participants) | 2033
  9 months | 0 [0 to 2.2]
  10 months: number analyzed (Participants) | 2032
  10 months | 0.6 [0 to 3.3]
  11 months: number analyzed (Participants) | 2025
  11 months | 0.7 [0 to 3.7]

ADVERSE EVENTS:
Time Frame: No AEs or SAEs were reported in this study.
Description: The study does not include the administration of any vaccine and no AEs or SAEs were reported in this study. Pregnancy outcomes and events of interests reported in the record did not meet the criteria for AEs or SAEs according to the standard definition in the protocol. Deaths reported in the all-cause mortality module include neonatal deaths, infant deaths and maternal deaths, while deaths reported in the participant flow include only infant deaths.
Arm/Group | Pregnant Women/Mothers Group | Neonates/Infants Group
All-Cause Mortality (participants affected / at risk) | 1/2311 | 23/2181
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study period partly overlapped with COVID-19 pandemic. RSV LRTI findings might not reflect a standard RSV season due to low virus circulation, social distancing, travel restriction and other actions to control COVID-19 spreading. GAIA classification is not used as care standard in participating sites. Some sites might face challenges into classify the outcomes of interest. Background rates for less frequent events were difficult to estimate due to the relatively limited size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03614676/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03614676/SAP_001.pdf